CLINICAL TRIAL: NCT01519700
Title: A Randomized, Double-blind, Parallel-group, Multi-center Phase III Study Comparing the Efficacy and Safety of EP2006 and Neupogen® in Breast Cancer Patients Treated With Myelosuppressive Chemotherapy
Brief Title: Phase III Study Comparing the Efficacy and Safety of EP2006 and Filgrastim
Acronym: PIONEER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EP06-302; 2010-024481-22 (EudraCT Number)
Record Dates: First submitted 2012-01-13; First posted 2012-01-27 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Chemotherapy Associated Neutropenia; Breast Cancer
Keywords: Filgrastim; G-CSF, neutropenia; supportive care; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EP2006 (Experimental): Eligible patients will be teated with EP2006
  Interventions: Drug: EP2006
- Filgrastim (Active Comparator): Eligible patients will be teated with Filgrastim
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: EP2006 — Eligible patients will be teated with EP2006
  Other Names: Filgrastim
  Arms: EP2006
Drug: Filgrastim — Eligible patients will be teated with Filgrastim
  Arms: Filgrastim

SUMMARY:
The study will assess the efficacy of EP2006 compared to Filgrastim with respect to the mean duration of severe neutropenia during treatment with myelosuppressive chemotherapy in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven breast cancer, eligible for neoadjuvant or adjuvant myelosuppressive chemotherapy
2. Women ≥ 18 years of age
3. Estimated life expectancy of more than six months

Exclusion Criteria:

1. Previous or concurrent malignancy except non-invasive non-melanoma skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least ten years prior to study entry
2. Any serious illness or medical condition that may interfere with safety, compliance, response to the products under investigation and their evaluation, e.g.:

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Chair — Sandoz
Locations (26):
- Insitut Onkologie a Rehabilitaca na Plesi, Ves Pod Plesi 110, Czechia
- Hungary (6):
  - Semmelweis Egyetem, III. Belgyogyaszati Klinika, Budapest
  - Fovarosi Onkormanyzat Uzsoki utcai Korhaz, Onkoradiologia, Budapest
  - DE OEC, Onkologiai Tanszek, Debrecen
  - Josa Andras Oktato Korhaz Nonprofit Kft, Nyíregyháza
  - Fejer Megyei Szent Gyorgy Korhaz, Onkologiai Osztaly, Székesfehérvár
  - Vas Megyei Markusovszky Korhaz, Onkoradiologiai Osztaly, Szombathely
- Daugavpils Regional Hospital, Daugavpils, Latvia
- Russia (11):
  - Institution of the Russian Academy of Medical Sciences Medical Radiology Research Center RAMS, Moscow, Krasnogorsk District
  - State Healthcare Institution (SHI) "Leningrad Regional Oncological Dispensary" at the Surgery Department 2, Kuzmolovsky, Leningradskaya Oblast'
  - State Medical-Prophylactic Institution SMPI Reginal Clinical Oncological Dispensary, Chelyabinsk
  - State Healthcare Institution (SHI) "Clinical Oncological Dispensary №1" of Healthcare Department of Krasnodar Territory, Krasnodar
  - Institution of the Russian Academy of Medical Sciences Russian Oncology Research Center n.a. N.N.Blochin of RAMS", Surgery Department of the Female Reproductive System Tumors, Moscow
  - Affiliate No1 of State Healthcare Institution (SHI) "Nizhny Novgorod Regional Oncological Dispensary", Nizhny Novgorod
  - Institution of the Russian Academy of Medical Sciences Medical Radiology Research Center RAMS, Obninsk
  - State Healthcare Institution SHI Pyatigorsk Oncological Dispensary, Pyatigorsk
  - Non-State Healthcare Institution NSHI, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution (SPb SHI) "City Clinical Oncological Dispensary", Saint Petersburg
  - State Healthcare Institution (SHI)"Voronezh Regional Clinical Oncological Dispensary", Voronezh
- Fakultna nemocnica Nitra, Oddelenie radioterapie a klinickej onkologie, Nitra, Slovakia
- Ukraine (6):
  - Communal Institution "Krivorizhskiy oncology dispensary" of Dnipropetrovsk regional Council, Chemotherapy Department, Kryvyi Rih, Dnipropetrovsk Oblast
  - Communal Institution "Dnipropetrovsk Сity multiple-discipline Clinical Hospital 4" of Dnipropetrovsk Regional Council, Dnipropetrovsk
  - Medical center of Limited Liability Company "Inter", Luhansk
  - Lviv state oncological regional treatment-and-diagnostics center, Chemotherapy Department, Lviv
  - Communal Institution "Odesa regional clinical hospital", Mammology Center, Odesa
  - Vinnytsya Regional Clinical Oncological Center, Chemotherapy Department, Vinnitsya

REFERENCES:
- [Derived] Blackwell K, Semiglazov V, Krasnozhon D, Davidenko I, Nelyubina L, Nakov R, Stiegler G, Singh P, Schwebig A, Kramer S, Harbeck N. Comparison of EP2006, a filgrastim biosimilar, to the reference: a phase III, randomized, double-blind clinical study in the prevention of severe neutropenia in patients with breast cancer receiving myelosuppressive chemotherapy. Ann Oncol. 2015 Sep;26(9):1948-1953. doi: 10.1093/annonc/mdv281. Epub 2015 Jun 28. PMID 26122726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of women of 18 years or older with histologically proven breast cancer who were eligible for neoadjuvant or adjuvant treatment with TAC chemotherapy. The study was aimed to randomize a total of 192 patients in approximately 65 centers worldwide.
Pre-assignment Details: The study started with a screening period of up to 21 days. During the screening period, the eligibility of the patients to participate in the study was assessed based on safety evaluations. After completion of the screening period, the patients were randomized to either EP2006 or US-licensed Neupogen® in four groups (see below).
Groups:
- EP2006: Patients remained on EP2006 (their initial treatment) throughout the study daily dose of 5 mcg/kg body weight, subcutaneously
- EP2006 + Neupogen: Patients received alternating treatment with EP2006 or Neupogen starting with the second cycle, daily dose of 5 mcg/kg body weight, subcutaneously
- Neupogen + EP2006: Patients received alternating treatment with Neupogen or EP2006 starting with the 2nd cycle, daily dose of 5 mcg/kg body weight, subcutaneously
- Neupogen: Patients remained on Neupogen (their initial treatment) throughout the study, daily dose of 5 mcg/kg body weight, subcutaneously
Period: Overall Study
Arm/Group | EP2006 | EP2006 + Neupogen | Neupogen + EP2006 | Neupogen
Started | 54 | 55 | 55 | 54
Treated Cycle 1 EP2006 | 53 | 54 | 0 | 0
Treated Cycle 1 Neupogen | 0 | 0 | 55 | 52
Treated Cycle 2 EP2006 | 52 | 0 | 55 | 0
Treated Cycle 2 Neupogen | 0 | 52 | 0 | 51
Treated Cycle 3 EP2006 | 51 | 51 | 0 | 0
Treated Cycle 3 Neupogen | 0 | 0 | 54 | 51
Treated Cycle 4 EP2006 | 51 | 0 | 50 | 0
Treated Cycle 4 Neupogen | 0 | 51 | 0 | 50
Treated Cycle 5 EP2006 | 46 | 49 | 0 | 0
Treated Cycle 5 Neupogen | 0 | 0 | 48 | 50
Treated Cycle 6 EP2006 | 45 | 0 | 48 | 0
Treated Cycle 6 Neupogen | 0 | 49 | 0 | 49
Completed | 45 | 49 | 48 | 47
Not Completed | 9 | 6 | 7 | 7
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 3 | 2
Not completed — Other Reason | 2 | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The safety set consists of all patients who received at least one dose of study drug and had at least one post-baseline safety assessment
Groups:
- EP2006: Patients remained on EP2006 (their initial treatment) throughout the study
- EP2006 + Neupogen: Patients received alternating treatment with EP2006 or Neupogen starting with the second cycle
- Neupogen + EP2006: Patients received alternating treatment with Neupogen or EP2006 starting with the 2nd cycle
- Neupogen: Patients remained on Neupogen (their initial treatment) throughout the study
- Total: Total of all reporting groups
Arm/Group | EP2006 | EP2006 + Neupogen | Neupogen + EP2006 | Neupogen | Total
Number analyzed (Participants) | 53 | 54 | 55 | 52 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (11.16) | 47.5 (11.64) | 49.7 (11.05) | 46.9 (10.91) | 48.9 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 55 | 52 | 214
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Grade 4 Neutropenia During Cycle 1 of Chemotherapy
Description: Mean duration of severe neutropenia, defined as the mean number of consecutive days with Grade 4 neutropenia (ANC less than 0.5*10^9 cells/L)
Time Frame: 21 days (Cycle 1 of chemotherapy treatment)
Population: PP population
Measure: Mean (Standard Deviation); unit: Days
Groups:
- EP2006 + EP2006 & Neupogen: All subjects randomized to receive either EP2006 in Cycle 1
- Neupogen + Neupogen & EP2006: All subjects randomized to receive Neupogen in Cycle 1
Arm/Group | EP2006 + EP2006 & Neupogen | Neupogen + Neupogen & EP2006
Number analyzed (Participants) | 101 | 103
Days | 1.17 (1.11) | 1.2 (1.02)
Statistical Analysis 1: Comparison: EP2006 + EP2006 & Neupogen; Test type: Non-Inferiority or Equivalence — Non-inferiority limit: -1 day Power: 90% Confidence level: 97.5% Randomization ratio: 1:1 (EP2006:Neupogen); Mean Difference (Net) = 0.04, 97.5% CI 1-sided [lower limit -0.26] — The one-sided 97.5% Confidence Interval: [-0.26, ∞)

2. Secondary Outcome: Incidence of Febrile Neutropenia
Description: Incidence of febrile neutropenia by duraton within each cycle and across all cycles. Febrile neutropenia is defined as oral temperature greater than or equal 38.3°C while having an Absolute Neutrophil Count < 0.5*10^9 cells/L (both measured on the same day)
Time Frame: 21 weeks/ 6 cycles
Population: SAF-I (alternating safety) set: patients who received at least one dose of study medication after Cycle 1.
Measure: Number; unit: participants
Groups:
- Total: All patients
Arm/Group | EP2006 | EP2006 + Neupogen | Neupogen + EP2006 | Neupogen | Total
Number analyzed (Participants) | 52 | 52 | 55 | 51 | 210
participants
  Cycle 1 - 0 Days duration | 50 | 49 | 54 | 51 | 204
  Cycle 1 - 1 Day duration | 2 | 3 | 0 | 0 | 5
  Cycle 1 - 2 Days duration | 0 | 0 | 1 | 0 | 1
  Cycle 2 - 0 Days duration | 52 | 51 | 55 | 51 | 209
  Cycle 2 - 1 Day duration | 0 | 1 | 0 | 0 | 1
  Cycle 3 - 0 Days duration | 51 | 51 | 54 | 51 | 207
  Cycle 4 - 0 Days duration | 51 | 51 | 50 | 50 | 202
  Cycle 5 - 0 Days duration | 45 | 48 | 48 | 50 | 191
  Cycle 5 - 1 Day duration | 0 | 1 | 0 | 0 | 1
  Cycle 6 - 0 Days duration | 43 | 48 | 48 | 49 | 188
  Cycle 6 - 1 Day duration | 1 | 1 | 0 | 0 | 2
  All Cycles - 0 Days duration | 49 | 46 | 54 | 51 | 200
  All Cycles - 1 Day duration | 3 | 6 | 0 | 0 | 9
  All Cycles - 2 Days duration | 0 | 0 | 1 | 0 | 1

3. Secondary Outcome: Number of Days of Fever
Description: Number of days of fever by cycle. Fever is defined as oral temperature greater than or equal to 38.3°C.
Time Frame: 21 weeks/ 6 cycles
Population: PP-I (alternating Per-Protocol) set: randomized patients who completed all six chemotherapy cycles without major protocol violations.
Measure: Number; unit: participants
Arm/Group | EP2006 | EP2006 + Neupogen | Neupogen + EP2006 | Neupogen | Total
Number analyzed (Participants) | 40 | 45 | 44 | 46 | 175
participants
  Cycle 1 - No | 39 | 41 | 42 | 46 | 168
  Cycle 1 - Yes | 1 | 4 | 2 | 0 | 7
  Cycle 2 - No | 36 | 43 | 44 | 46 | 169
  Cycle 2 - Yes | 4 | 2 | 0 | 0 | 6
  Cycle 3 - No | 40 | 44 | 44 | 45 | 173
  Cycle 3 - Yes | 0 | 1 | 0 | 1 | 2
  Cycle 4 - No | 40 | 44 | 43 | 46 | 173
  Cycle 4 - Yes | 0 | 1 | 1 | 0 | 2
  Cycle 5 - No | 40 | 44 | 43 | 45 | 172
  Cycle 5 - Yes | 0 | 1 | 1 | 1 | 3
  Cycle 6 - No | 39 | 44 | 44 | 46 | 173
  Cycle 6 - Yes | 1 | 1 | 0 | 0 | 2

4. Secondary Outcome: Depth of Absolute Neutrophil Count Nadir
Description: Depth of Absolute Neutrophil Count Nadir, defined as the patient's lowest Absolute Neutrophil Count in cycle 1
Time Frame: Cycle 1/ 21 days
Population: FAS (full analysis) set: all patients who received at least one dose of study medication, analyzed according to randomization allocation
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Groups:
- Total: All patients in Cycle 1
Arm/Group | EP2006 + EP2006 & Neupogen | Neupogen + Neupogen & EP2006 | Total
Number analyzed (Participants) | 107 | 107 | 214
10^9 cells/L | 0.808 (1.3694) | 0.744 (1.2906) | 0.776 (1.3278)

5. Secondary Outcome: Time to Absolute Neutrophil Count Recovery
Description: Time to Absolute Neutrophil Count recovery, defined as the time in days from Absolute Neutrophil Count nadir until the patient's Absolute Neutrophil Count increases to more or equal to 2*10^9 cells/L after the nadir in cycle 1
Time Frame: Cycle 1/ 21 days
Population: FAS (full analysis) set: all patients who received at least one dose of study medication, analyzed according to randomization allocation. In the EP2006 + EP2006 & Neupogen group, one patient's time to Absolute Neutrophil Count recovery could not be measured as the nadir was the last measured timepoint.
Measure: Median (Full Range); unit: Days
Arm/Group | EP2006 + EP2006 & Neupogen | Neupogen + Neupogen & EP2006 | Total
Number analyzed (Participants) | 106 | 107 | 213
Days | 2.0 [0 to 6] | 2.0 [0 to 4] | 2.0 [0 to 6]

6. Secondary Outcome: Frequency of Infections
Description: Frequency of infections by cycle and across all cycles
Time Frame: 21 Weeks/ 6 cycles
Population: SAF-I (alternating safety) set: patients who received at least one dose of study medication after Cycle 1. Comparison made for alternating versus non-alternating treatment groups.
Measure: Number; unit: participants
Groups:
- EP2006 + Neupogen: All subjects randomized to receive either EP2006 or Neupogen.
- EP2006 & Neupogen + Neupogen & EP2006: All subjects randomized to receive EP2006 & Neupogen + Neupogen & EP2006.
Arm/Group | EP2006 + Neupogen | EP2006 & Neupogen + Neupogen & EP2006 | Total
Number analyzed (Participants) | 103 | 107 | 210
participants
  Cycle 1 - No | 102 | 104 | 206
  Cycle 1 - Yes | 1 | 3 | 4
  Cycle 2 - No | 100 | 102 | 202
  Cycle 2 - Yes | 3 | 5 | 8
  Cycle 3 - No | 102 | 107 | 209
  Cycle 3 - Yes | 1 | 0 | 1
  Cycle 4 - No | 101 | 104 | 205
  Cycle 4 - Yes | 2 | 3 | 5
  Cycle 5 - No | 101 | 106 | 207
  Cycle 5 - Yes | 2 | 1 | 3
  Cycle 6 - No | 102 | 106 | 208
  Cycle 6 - Yes | 1 | 1 | 2
  All Cycles - No | 96 | 97 | 193
  All Cycles - Yes | 7 | 10 | 17

7. Secondary Outcome: Incidence of Hospitalizations Due to Febrile Neutropenia
Description: Incidence of hospitalizations due to Febrile Neutropenia
Time Frame: 21 Weeks/ 6 cycles
Population: SAF-I (alternating safety) set: patients who received at least one dose of study medication after Cycle 1.
Measure: Number; unit: participants
Arm/Group | EP2006 | EP2006 + Neupogen | Neupogen + EP2006 | Neupogen | Total
Number analyzed (Participants) | 52 | 52 | 55 | 51 | 210
participants
  No | 50 | 50 | 55 | 51 | 206
  Yes | 2 | 1 | 0 | 1 | 4

ADVERSE EVENTS:
Arm/Group | EP2006 | EP2006 + Neupogen | Neupogen + EP2006 | Neupogen
Serious Adverse Events (participants affected / at risk) | 6/53 | 4/54 | 1/55 | 3/52
Other Adverse Events (participants affected / at risk) | 50/53 | 51/54 | 52/55 | 50/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP2006 (N=53) | EP2006 + Neupogen (N=54) | Neupogen + EP2006 (N=55) | Neupogen (N=52)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP2006 (N=53) | EP2006 + Neupogen (N=54) | Neupogen + EP2006 (N=55) | Neupogen (N=52)
Alopecia (Skin and subcutaneous tissue disorders) | 41 (43) | 44 (45) | 43 (46) | 43 (44)
Erythema (Skin and subcutaneous tissue disorders) | 5 (15) | 2 (3) | 6 (19) | 6 (23)
Asthenia (General disorders) | 20 (66) | 28 (98) | 32 (111) | 28 (101)
Fatigue (General disorders) | 17 (52) | 9 (17) | 11 (38) | 13 (38)
Hypothermia (General disorders) | 0 (0) | 3 (6) | 1 (14) | 1 (1)
Pyrexia (General disorders) | 6 (9) | 3 (8) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 29 (103) | 33 (95) | 32 (116) | 37 (149)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 11 (14) | 13 (21) | 8 (11)
Vomiting (Gastrointestinal disorders) | 9 (27) | 10 (22) | 10 (21) | 9 (19)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 5 (10) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (8) | 2 (2) | 4 (7) | 3 (6)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (33) | 20 (46) | 19 (60) | 19 (60)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (8) | 4 (4) | 6 (8) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (4) | 3 (5) | 3 (4)
Musculosceletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (2) | 2 (3) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (21) | 7 (18) | 6 (20) | 6 (22)
Anaemia (Blood and lymphatic system disorders) | 6 (10) | 5 (9) | 4 (6) | 11 (24)
Leucopenia (Blood and lymphatic system disorders) | 4 (21) | 4 (12) | 2 (3) | 3 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (8) | 0 (0) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (6) | 3 (3) | 2 (2) | 1 (1)
Periferal sensory neur. (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 8 (21) | 4 (8) | 3 (6) | 13 (32)
Flushing (Vascular disorders) | 1 (3) | 3 (10) | 0 (0) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall provide Sponsor with any presentation at least 15 working days prior to disclosure and any other publication at least 45 working days prior to disclosure. Sponsor may require amendments on reasonable grounds: (a) accuracy of publication; (b) confidentiality of proprietary information; (c) intellectual property protection; (d) to enable further information to be provided. Sponsor may require publications or presentations to be delayed up to four (4) months to enable patent application.